CLINICAL TRIAL: NCT00109356
Title: A Phase 1/2, Open Label, Dose Escalation Study of AQ4N for Safety, Tolerability, Pharmacokinetics and Activity in Patients With Lymphoid Neoplasms
Brief Title: Study of AQ4N in Patients With Non Hodgkin's Lymphoma, Chronic Lymphocytic Leukemia, or Small Lymphocytic Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Novacea (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 021-002
Record Dates: First submitted 2005-04-27; First posted 2005-04-27 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia
Keywords: Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — AQ4N; Drug Therapy

INTERVENTIONS:
Drug: AQ4N (Chemotherapy)

SUMMARY:
The purpose of this study is to find answers to the following questions:

* What is the largest dose of AQ4N that can be given safely one time every three weeks for 24 weeks?
* What are the side effects of AQ4N when given according to this schedule?
* How much AQ4N is in the blood at certain times after administration and how does the body get rid of the drug?
* Will AQ4N help treat lymphoid cancer?

DETAILED DESCRIPTION:
All patients in this study will receive AQ4N one time every three weeks for a maximum of 24 weeks. Each patient will receive the same dose for the entire time he/she is on the study. However, some patients may receive a different dose than other patients depending upon when they enter the study.

When the study begins, the first three patients will receive a dose of 400 mg/m2. After they have all been observed for 2 weeks, and if side effects do not occur or are tolerable, another three patients will enter the study at a higher dose. The increase in dose may continue with new patient groups until side effects reach a point where they are not tolerated. At that point no higher doses will be tried and more patients will be allowed to enter at one or two lower doses where the side effects were tolerated.

Up to 55 patients will be entered in this study at up to 8 research centers in the United States. Study duration will be approximately 27 weeks or 8 treatment cycles (One treatment cycle lasts 3 weeks and begins on Day 1 with an infusion of AQ4N.)

The following procedures will be completed at the time of screening and throughout the study: review of medical and cancer history, previous cancer treatments, and current medications, a complete physical exam, and blood (4 to 6 teaspoons) and urine tests. Two additional tests to evaluate the heart, an electrocardiogram (ECG) and a multiple gated acquisition assessment (MUGA) will be performed. Cancer progression will be monitored by a computed tomography scan (CT scan) and a bone marrow biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Non-Hodgkin's Lymphoma, Chronic Lymphocytic Leukemia, or Small Lymphocytic Leukemia
* Tumor specimen available for evaluation (please provide 10 unstained slides)
* Relapse after receiving primary treatment and at least one salvage therapy
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Laboratory test measurements
* Females of childbearing potential must have a negative pregnancy test result within 3 days prior to the first dose and must agree to use an effective contraceptive method during the course of the study and for 6 months following the last dose of study drug.
* Older than 18 years of age
* Available for periodic blood sampling

Exclusion Criteria:

* Certain cardiac problems
* Previous donor stem cell transplant
* Known HIV, Hepatitis B, Hepatitis C infection
* Previous chemotherapy, radiation or other investigational drug treatments within 4 weeks of first planned dose of study drug
* Major surgery within four weeks of first planned dose of study drug
* Any active viral, bacterial, or fungal infection within four weeks of first planned dose of study drug
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Start 2005-03; Study Completion 2007-03

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Response duration and time to tumor progression
Time to treatment failure
Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Medical College of Cornell University/ New York Presbyterian Hospital, New York, New York, United States